CLINICAL TRIAL: NCT02390050
Title: A Phase 2b, Multi-center, Double-blind, Placebo-controlled, Dose Range Finding Study to Evaluate the Effect of Bexagliflozin Tablets on HbA1c in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Dose Range Finding Study to Evaluate the Effect of Bexagliflozin Tablets in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-449
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bexagliflozin tablets, 5 mg (Active Comparator): Bexagliflozin tablets, 5 mg, once daily by mouth before breakfast
  Interventions: Drug: Bexagliflozin tablets
- Bexagliflozin tablets, 10 mg (Active Comparator): Bexagliflozin tablets, 10 mg, once daily by mouth before breakfast
  Interventions: Drug: Bexagliflozin tablets
- Bexagliflozin tablets, 20 mg (Active Comparator): Bexagliflozin tablets, 20 mg, once daily by mouth before breakfast
  Interventions: Drug: Bexagliflozin tablets
- Bexagliflozin tablets, placebo (Placebo Comparator): Bexagliflozin tablets, placebo, once daily by mouth before breakfast
  Interventions: Drug: Bexagliflozin tablets, placebo

INTERVENTIONS:
Drug: Bexagliflozin tablets — Bexagliflozin tablets are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
  Other Names: Code name: EGT0001442
  Arms: Bexagliflozin tablets, 10 mg; Bexagliflozin tablets, 20 mg; Bexagliflozin tablets, 5 mg
Drug: Bexagliflozin tablets, placebo — Bexagliflozin tablets, placebo, are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
  Arms: Bexagliflozin tablets, placebo

SUMMARY:
The purpose of this study was to investigate the effect of bexagliflozin in lowering hemoglobin A1c (HbA1c) levels in patients with type 2 diabetes mellitus (T2DM). Bexagliflozin is an orally administered drug for the treatment of T2DM and is classified as a Sodium Glucose co-Transporter 2 (SGLT2) Inhibitor. This study was to enroll both treatment naive and those subjects previously treated with one oral hypoglycemic agent (OHA). Approximately 320 subjects eligible for randomization was to receive bexagliflozin tablets, 5, 10, 20 mg or placebo, once daily for 12 weeks in an outpatient setting.

DETAILED DESCRIPTION:
The study was a phase 2b multicenter, double-blind, placebo-controlled parallel group study to assess the effect of once daily bexagliflozin tablets on HbA1c in either treatment-naïve T2DM subjects or in subjects who were treated with one oral anti-diabetic agent. Treatment naïve subjects were eligible if their HbA1c values were between 7% and 8.5% at the screening visit while subjects who were treated with one oral hypoglycemic agent (OHA) were eligible if their HbA1c value was between 6.5% and 8.5% at screening and underwent a 6 or 10 week washout period. In addition, all eligible subjects underwent a two week placebo run-in period and those who showed good compliance in taking study medication (i.e., missed no more than one dose during the run-in period) during this period and whose HbA1c values were between 7 and 8.5% at the end of the run-in period were eligible for randomization.

ELIGIBILITY:
The following subjects were eligible for randomization:

1. men or women ≥ 20 years of age at screening. Women of childbearing potential must test negative by urine pregnancy test.
2. were treatment naïve or taking one oral anti-diabetic medication in combination with diet and exercise
3. were diagnosed with T2DM with HbA1c levels at screening between 7.0% and 8.5% (inclusive) if treatment naïve or with HbA1c levels between 6.5 and 8.5% (inclusive) if on one oral anti-diabetic medication
4. had a body mass index (BMI) ≤ 40 kg/m2
5. were taking stable doses of medication for hypertension or hyperlipidemia that has not changed for at least 30 days prior to screening (if applicable)
6. were able to comprehend the study participation requirements and willing to provide written informed consent in accordance with institutional and regulatory guidelines
7. were able to maintain adequate glycemic control at the run-in visit (for subjects who complete the washout)
8. had an HbA1c between 7.0 and 8.5% (inclusive) prior to randomization (day -3 to -5)
9. were capable of adhering to the investigational product administration requirements as evidenced by omission of no more than one dose of run-in medication

Subjects who exhibited any of the following characteristics were to be ineligible for randomization:

1. Diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young
2. Used parenteral therapy for treatment of diabetes
3. Pregnancy or current breastfeeding status
4. Hemoglobinopathy or carrier status for hemoglobin alleles that affect HbA1c measurement
5. Genitourinary tract infection within 6 weeks of screening or history of ≥3 genitourinary infections requiring treatment within 6 months of screening
6. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 at screening.
7. Uncontrolled hypertension at screening
8. A positive result on hepatitis B surface antigen, hepatitis C, or positive result from screen for drugs of abuse
9. History of human immunodeficiency virus infection
10. Life expectancy < 2 years
11. History of New York Heart Association Class 4 heart failure within 3 months of screening
12. History of myocardial infarction, unstable angina, stroke, or hospitalization for heart failure within 3 months of screening
13. History of treatment with an investigational drug within 30 days or within 7 half lives of the investigational drug, whichever is longer
14. Previous treatment with bexagliflozin
15. Had taken or within 6 months of taking any Sodium Glucose Transporter 2 (SGLT2) inhibitors prior to screening
16. Participation of another interventional trial
17. Not able to comply with the study scheduled visits
18. Affected by any condition, disease, disorder, or clinically relevant abnormality that, in the opinion of the investigator, would jeopardize the subject's appropriate participation in this study.
19. Liver function tests resulting in Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 2.5 x upper limit of normal (ULN) or total bilirubin ≥ 1.5 x ULN, with the exception of isolated Gilbert's syndrome ,at screening
20. Exhibited fasting plasma glucose ≥ 250 mg/dL (13.9 mmol/L) on two or more consecutive days prior to randomization or exhibited severe clinical signs or symptoms of hyperglycemia during the washout or run-in periods, including weight loss, blurred vision, increased thirst, or increased urination, or fatigue
21. Fasting Plasma Glucose ≥ 250 mg/dL at randomization
22. Prior renal transplantation or evidence of nephrotic syndrome, defined as a urine albumin-to-creatinine ratio (UACR) > 2000 mg/g at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Paul Lock, M.D., Study Director — Theracos
Locations (50):
- United States (32):
  - Phoenix Medical Research Institute LLC, Peoria, Arizona
  - Advanced Arizona Clinical Research, Tucson, Arizona
  - Hope Clinical Research, LLC, Canoga Park, California
  - Catalina Research Institute, Chino, California
  - National Research Institute, Huntington Park, California
  - Long Beach Clinical Trials, Long Beach, California
  - Synergy San Diego, National City, California
  - Northern California Research, Sacramento, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Infosphere Clinical Research, Inc, West Hills, California
  - M&O Clinical Research LLC, Fort Lauderdale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Compass Research North, Leesburg, Florida
  - Sweet Hope Research Specialty, Inc, Miami Lakes, Florida
  - Sunshine Research Center, Opa-locka, Florida
  - Compass Research LLC, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - PICR Clinic, Atlanta, Georgia
  - Sundance Clinical Research, St Louis, Missouri
  - Premier Research Ltd, Trenton, New Jersey
  - Regional Clinical Research, Inc, Endwell, New York
  - Calabash Medical Center, Calabash, North Carolina
  - Diabetes & Endocrinology Consultants PC, Morehead City, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - CTI Research, Cincinnati, Ohio
  - Summit Research Group, LLC, Stow, Ohio
  - Columbia Research Group, Inc., Portland, Oregon
  - Detweiler Family Medicine and Associate, P.C., Lansdale, Pennsylvania
  - North Myrtle Beach Family Practice, Myrtle Beach, South Carolina
  - Global Medical Research, DeSoto, Texas
  - Rockwood Medical Clinic, Fort Worth, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
- Japan (18):
  - Medical Corporation Hitomi-kai Motomachi Takatsuka Naika Clinic, Yokohama Naka-ku, Kanagawa
  - Medical Corporation Hayashi katagihara Clinic, Nishikyo-ku, Kyoto
  - Medical Corporation KEISEIKAI Kajiyama clinic, Ukyou-ku, Kyoto
  - Ikeoka Medical Corp. Ikeoka Clinic, Joto-ku, Osaka
  - Miyauchi Medical Center, Takatsuki-shi, Osaka
  - Medical Corporation Senrichuo Ekimae Clinic, Toyonaka-shi, Osaka
  - Medical Corporation Segawa Hospital, Hikigun Ogawamachi, Saitama
  - Medical Corporation Yukeikai Asano Clinic, Kawagoe-shi, Saitama
  - Medical Corporation Ishii Internal Medicine Clinic, Kawaguchi, Saitama
  - Medical Corporation Fusanokai Shimizu Clinic Fusa, Saitama-shi, Saitama
  - Medical Corp. SEIKOUKAI New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Medical Corporation Jototowakai Shinkoiwa ekimae sogo Clinic, Katsushika-ku, Tokyo
  - Medical Corporation IHL Pedi Shiodome Medical Clinic, Minato-ku, Tokyo
  - Medical Corporation IHL Shinagawa East One Medical Clinic, Minato-ku, Tokyo
  - Kenkokan Suzuki Clinic, Ōta-ku, Tokyo
  - Medical Corporation Souyu-kai Hirahata Clinic, Shibuya-ku, Tokyo
  - Medical Corporation Yuhokai Miho-Clinic, Shinagawa-ku, Tokyo
  - Ikebukuro Metropolitan Clinic, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Background] Matsuo S, Imai E, Horio M, Yasuda Y, Tomita K, Nitta K, Yamagata K, Tomino Y, Yokoyama H, Hishida A; Collaborators developing the Japanese equation for estimated GFR. Revised equations for estimated GFR from serum creatinine in Japan. Am J Kidney Dis. 2009 Jun;53(6):982-92. doi: 10.1053/j.ajkd.2008.12.034. Epub 2009 Apr 1. PMID 19339088
- [Background] National Research Council (US) Panel on Handling Missing Data in Clinical Trials. The Prevention and Treatment of Missing Data in Clinical Trials. Washington (DC): National Academies Press (US); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK209904/ PMID 24983040
- [Background] Palaniappan LP, Wong EC, Shin JJ, Fortmann SP, Lauderdale DS. Asian Americans have greater prevalence of metabolic syndrome despite lower body mass index. Int J Obes (Lond). 2011 Mar;35(3):393-400. doi: 10.1038/ijo.2010.152. Epub 2010 Aug 3. PMID 20680014
- [Background] Santer R, Kinner M, Lassen CL, Schneppenheim R, Eggert P, Bald M, Brodehl J, Daschner M, Ehrich JH, Kemper M, Li Volti S, Neuhaus T, Skovby F, Swift PG, Schaub J, Klaerke D. Molecular analysis of the SGLT2 gene in patients with renal glucosuria. J Am Soc Nephrol. 2003 Nov;14(11):2873-82. doi: 10.1097/01.asn.0000092790.89332.d2. PMID 14569097
- [Background] Scheen AJ, Van Gaal LF. Combating the dual burden: therapeutic targeting of common pathways in obesity and type 2 diabetes. Lancet Diabetes Endocrinol. 2014 Nov;2(11):911-22. doi: 10.1016/S2213-8587(14)70004-X. Epub 2014 Feb 19. PMID 24731666
- [Background] Schwartz S, Fabricatore AN, Diamond A. Weight reduction in diabetes. Adv Exp Med Biol. 2012;771:438-58. doi: 10.1007/978-1-4614-5441-0_31. PMID 23393695
- [Background] van den Heuvel LP, Assink K, Willemsen M, Monnens L. Autosomal recessive renal glucosuria attributable to a mutation in the sodium glucose cotransporter (SGLT2). Hum Genet. 2002 Dec;111(6):544-7. doi: 10.1007/s00439-002-0820-5. Epub 2002 Sep 27. PMID 12436245
- [Background] Japan Diabetes Society (2012). Treatment Guidance for Diabetes 2012-2013.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet once daily before breakfast
  Placebo tablets are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
- Bexagliflozin 5 mg: Bexagliflozin tablet, 5 mg, once daily before breakfast
  Bexagliflozin tablets are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
- Bexagliflozin 10 mg: Bexagliflozin tablet, 10 mg, once daily before breakfast
  Bexagliflozin tablets are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
- Bexagliflozin 20 mg: Bexagliflozin tablet, 20 mg, once daily before breakfast
  Bexagliflozin tablets are blue caplet-shaped, film-coated tablets that are intended for use in investigational studies in humans.
Period: Overall Study
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Started | 72 | 72 | 72 | 76
Completed | 65 | 67 | 68 | 69
Not Completed | 7 | 5 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg | Total
Number analyzed (Participants) | 72 | 72 | 72 | 76 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.42) | 59.0 (10.22) | 59.4 (8.99) | 59.5 (10.81) | 59.2 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 31 | 26 | 112
  Male | 42 | 47 | 41 | 50 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 12 | 15 | 58
  Not Hispanic or Latino | 57 | 55 | 58 | 61 | 231
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 37 | 38 | 39 | 41 | 155
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 9 | 8 | 30
  White | 27 | 27 | 23 | 26 | 103
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 33 | 37 | 142
  Japan | 36 | 36 | 39 | 39 | 150
Height [Mean (Standard Deviation); unit: cm] | 165.6 (10.63) | 165.7 (9.25) | 165.8 (9.03) | 166.0 (10.33) | 165.8 (9.79)
Body Weight [Mean (Standard Deviation); unit: kg] | 78.72 (19.747) | 80.52 (18.977) | 78.39 (17.589) | 78.84 (16.740) | 79.11 (18.204)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.54 (5.535) | 29.10 (5.211) | 28.35 (4.978) | 28.49 (5.010) | 28.62 (5.167)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c After 12 Weeks of Treatment
Description: Mixed model repeated measures (MMRM) analysis of covariance model (ANCOVA) with baseline HbA1c as a covariate will be fit to the available data, incorporating all visits at which HbA1c was measured for each subject including scheduled visits at Weeks 2, 6, and 12 as well as unscheduled visits for measurements of HbA1c. Treatment (placebo, 5 mg, 10 mg, 20 mg), study center, prior anti-diabetic treatment status, study visit and treatment-by-visit interaction will be applied as fixed effects and subject as a random effect. The least square mean (LSM) change from baseline to Week 12 was analyzed using the Mixed-Effect Model Repeated Measure (MMRM) Analysis of Covariance (ANCOVA) model using 95% Confidence Intervals (CIs) for the between-group mean changes.
Time Frame: 12 weeks
Population: Subjects who were randomized, took at least one dose of double-blind study medication, and had at least one post-randomization HbA1c measurement were included in the full analysis dataset (FAS). TheHbA1c change from baseline through 12 weeks, and the primary analysis is based on the available data and data obtained after rescue will be excluded and considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 64 | 65 | 68 | 68
percentage of glycated hemoglobin | 0.24 (0.08) | -0.31 (0.08) | -0.44 (0.08) | -0.56 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; Study center, treatment, visit and a treatment-by-visit interaction as fixed effects; prior anti-diabetic treatment and baseline HbA1c as covariates; Difference of LS Means = -0.55, 95% CI 2-sided [-0.76 to -0.34]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.68, 95% CI 2-sided [-0.89 to -0.47]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.80, 95% CI 2-sided [-1.01 to -0.59]

2. Secondary Outcome: Proportion of Subjects With HbA1c < 7%
Description: To assess the efficacy of bexagliflozin based on the proportion of subjects who reach the American Diabetes Associate (ADA) and the Japan Diabetes Society target HbA1c of <7%.
Time Frame: Baseline to up to 12 weeks
Population: Subjects with at least one post-baseline HbA1c value <7% met this endpoint. HbA1c values obtained after start of rescue medication were excluded from this analysis. The number and percentage of subjects with at least one HbA1c value <7% were summarized by treatment group for the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 72 | 71 | 72 | 75
Participants | 11 | 15 | 16 | 27
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Odds ratio of having at least 1 post-baseline HbA1c value <7% in the 5 mg bexagliflozin group was compared to placebo group; Test type: Superiority; p = 0.1308, Regression, Logistic; Treatment, country, baseline HbA1c and prior anti-diabetic treatment status as predictor variables and a dependable variable of 1 (<7%) or 0 (>7%); Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.8 to 5.3]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Odds ratio of having at least 1 post-baseline HbA1c value <7% in the 10 mg bexagliflozin group was compared to placebo group; Test type: Superiority; p = 0.1294, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.8 to 5.1]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Odds ratio of having at least 1 post-baseline HbA1c value <7% in the 20 mg bexagliflozin group was compared to placebo group; Test type: Superiority; p = 0.0015, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 4.2, 95% CI 2-sided [1.7 to 10.3]

3. Secondary Outcome: Change in Body Weight Over Time
Description: The body weight was analyzed on the full analysis set using the MMRM ANCOVA model used for the primary efficacy analysis.
Time Frame: Baseline to Week 2, Week 6 and Week 12
Population: Only subject with a value at the specified time is included
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 72 | 71 | 72 | 75
kg
  Week 2: number analyzed (Participants) | 71 | 71 | 72 | 75
  Week 2 | 0.00 (0.15) | -0.74 (0.16) | -0.76 (0.15) | -0.99 (0.15)
  Week 6: number analyzed (Participants) | 70 | 70 | 71 | 75
  Week 6 | 0.02 (0.19) | -1.00 (0.19) | -1.42 (0.19) | -1.49 (0.19)
  Week 12: number analyzed (Participants) | 69 | 69 | 71 | 69
  Week 12 | -0.14 (0.25) | -1.58 (0.25) | -1.72 (0.25) | -1.89 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Week 2: Difference in LS mean change in body weight from baseline to week 2 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.74, 95% CI 2-sided [-1.13 to -0.36]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Week 2: Difference in LS mean change in body weight from baseline to week 2 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.76, 95% CI 2-sided [-1.15 to -0.38]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Week 2: Difference in LS mean change in body weight from baseline to week 2 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.99, 95% CI 2-sided [-1.38 to -0.61]
Statistical Analysis 4: Comparison: Placebo vs Bexagliflozin 5 mg; Week 6: Difference in LS mean change in body weight from baseline to week 6 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.02, 95% CI 2-sided [-1.53 to -0.52]
Statistical Analysis 5: Comparison: Placebo vs Bexagliflozin 10 mg; Week 6: Difference in LS mean change in body weight from baseline to week 6 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.45, 95% CI 2-sided [-1.95 to -0.94]
Statistical Analysis 6: Comparison: Placebo vs Bexagliflozin 20 mg; Week 6: Difference in LS mean change in body weight from baseline to week 6 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.51, 95% CI 2-sided [-2.01 to -1.01]
Statistical Analysis 7: Comparison: Placebo vs Bexagliflozin 5 mg; Week 12: Difference in LS mean change in body weight from baseline to week 12 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; Study center, treatment, visit and a treatment-by-visit interaction as fixed effects; prior anti-diabetic treatment and baseline weight as covariates; Difference of LS Means = -1.44, 95% CI 2-sided [-2.12 to -0.76]
Statistical Analysis 8: Comparison: Placebo vs Bexagliflozin 10 mg; Week 12: Difference in LS mean change in body weight from baseline to week 12 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 3, analysis 7]; Difference of LS Means = -1.59, 95% CI 2-sided [-2.26 to -0.91]
Statistical Analysis 9: Comparison: Placebo vs Bexagliflozin 20 mg; Week 12: Difference in LS mean change in body weight from baseline to week 12 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 3, analysis 7]; Difference of LS Means = -1.75, 95% CI 2-sided [-2.43 to -1.08]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) Over Time
Description: The fasting plasma glucose (FPG) was analyzed on the full analysis set using the same MMRM ANCOVA model used in the primary efficacy analysis.
Time Frame: Baseline to Week 2, Week 6 and Week 12
Population: Only subject with a value at the specified time is included
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 72 | 71 | 72 | 75
mmol/L
  Week 2: number analyzed (Participants) | 71 | 71 | 72 | 75
  Week 2 | -0.07 (0.16) | -0.55 (0.16) | -0.97 (0.16) | -1.11 (0.15)
  Week 6: number analyzed (Participants) | 70 | 70 | 71 | 75
  Week 6 | 0.11 (0.17) | -0.82 (0.17) | -1.06 (0.17) | -0.99 (0.17)
  Week 12: number analyzed (Participants) | 69 | 69 | 71 | 69
  Week 12 | -0.11 (0.17) | -0.96 (0.17) | -1.16 (0.17) | -1.18 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Week 2: Difference in LS mean change in FPG from baseline to week 2 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.48, 95% CI 2-sided [-0.90 to -0.06]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Week 2: Difference in LS mean change in FPG from baseline to week 2 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.90, 95% CI 2-sided [-1.31 to -0.48]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Week 2: Difference in LS mean change in FPG from baseline to week 2 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.04, 95% CI 2-sided [-1.45 to -0.62]
Statistical Analysis 4: Comparison: Placebo vs Bexagliflozin 5 mg; Week 6: Difference in LS mean change in FPG from baseline to week 6 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.93, 95% CI 2-sided [-1.39 to -0.48]
Statistical Analysis 5: Comparison: Placebo vs Bexagliflozin 10 mg; Week 6: Difference in LS mean change in FPG from baseline to week 6 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.17, 95% CI 2-sided [-1.62 to -0.72]
Statistical Analysis 6: Comparison: Placebo vs Bexagliflozin 20 mg; Week 6: Difference in LS mean change in FPG from baseline to week 6 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.10, 95% CI 2-sided [-1.55 to -0.65]
Statistical Analysis 7: Comparison: Placebo vs Bexagliflozin 5 mg; Week 12: Difference in LS mean change in FPG from baseline to week 12 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; p = 0.0002, ANCOVA — P-value from Type III F-test; Study center, treatment, visit and a treatment-by-visit interaction as fixed effects; prior anti-diabetic treatment and baseline FPG as covariates; Difference of LS Means = -0.85, 95% CI 2-sided [-1.29 to -0.41]
Statistical Analysis 8: Comparison: Placebo vs Bexagliflozin 10 mg; Week 12: Difference in LS mean change in FPG from baseline to week 12 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 4, analysis 7]; Difference of LS Means = -1.05, 95% CI 2-sided [-1.49 to -0.60]
Statistical Analysis 9: Comparison: Placebo vs Bexagliflozin 20 mg; Week 12: Difference in LS mean change in FPG from baseline to week 12 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 4, analysis 7]; Difference of LS Means = -1.07, 95% CI 2-sided [-1.52 to -0.63]

5. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure Over Time
Description: The systolic blood pressure (SBP) and diastolic blood pressure (DBP) were analyzed on the full analysis set using the same MMRM ANCOVA model used in the primary efficacy analysis.
Time Frame: Baseline to Week 2, Week 6 and Week 12
Population: Only subject with a value at the specified time is included
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 72 | 71 | 72 | 75
mm Hg
  Week 2 SBP: number analyzed (Participants) | 71 | 71 | 72 | 75
  Week 2 SBP | -0.14 (1.42) | -0.33 (1.43) | -2.55 (1.42) | -4.39 (1.38)
  Week 2 DBP: number analyzed (Participants) | 71 | 71 | 72 | 75
  Week 2 DBP | 0.15 (0.89) | -0.03 (0.89) | -1.59 (0.88) | -2.00 (0.86)
  Week 6 SBP: number analyzed (Participants) | 70 | 70 | 71 | 75
  Week 6 SBP | -0.57 (1.44) | -1.40 (1.45) | -3.96 (1.44) | -3.07 (1.39)
  Week 6 DBP: number analyzed (Participants) | 70 | 70 | 71 | 75
  Week 6 DBP | -0.52 (0.92) | -0.27 (0.93) | -1.54 (0.92) | -0.36 (0.89)
  Week 12 SBP: number analyzed (Participants) | 69 | 69 | 71 | 69
  Week 12 SBP | 1.10 (1.56) | -1.06 (1.57) | -3.30 (1.55) | -2.73 (1.55)
  Week 12 DBP: number analyzed (Participants) | 69 | 69 | 71 | 69
  Week 12 DBP | 0.81 (0.95) | -1.43 (0.95) | -0.66 (0.94) | -1.23 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Week 2: Difference in LS mean change in SBP from baseline to week 2 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.19, 95% CI 2-sided [-3.90 to 3.51]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Week 2: Difference in LS mean change in SBP from baseline to week 2 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -2.41, 95% CI 2-sided [-6.09 to 1.28]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Week 2: Difference in LS mean change in SBP from baseline to week 2 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -4.25, 95% CI 2-sided [-7.93 to -0.58]
Statistical Analysis 4: Comparison: Placebo vs Bexagliflozin 5 mg; Week 2: Difference in LS mean change in DBP from baseline to week 2 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.18, 95% CI 2-sided [-2.50 to 2.13]
Statistical Analysis 5: Comparison: Placebo vs Bexagliflozin 10 mg; Week 2: Difference in LS mean change in DBP from baseline to week 2 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.74, 95% CI 2-sided [-4.03 to 0.56]
Statistical Analysis 6: Comparison: Placebo vs Bexagliflozin 20 mg; Week 2: Difference in LS mean change in DBP from baseline to week 2 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -2.15, 95% CI 2-sided [-4.45 to 0.14]
Statistical Analysis 7: Comparison: Placebo vs Bexagliflozin 5 mg; Week 6: Difference in LS mean change in SBP from baseline to week 6 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.84, 95% CI 2-sided [-4.57 to 2.90]
Statistical Analysis 8: Comparison: Placebo vs Bexagliflozin 10 mg; Week 6: Difference in LS mean change in SBP from baseline to week 6 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -3.39, 95% CI 2-sided [-7.12 to 0.34]
Statistical Analysis 9: Comparison: Placebo vs Bexagliflozin 20 mg; Week 6: Difference in LS mean change in SBP from baseline to week 6 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -2.51, 95% CI 2-sided [-6.21 to 1.20]
Statistical Analysis 10: Comparison: Placebo vs Bexagliflozin 5 mg; Week 6: Difference in LS mean change in DBP from baseline to week 6 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = 0.25, 95% CI 2-sided [-2.15 to 2.66]
Statistical Analysis 11: Comparison: Placebo vs Bexagliflozin 10 mg; Week 6: Difference in LS mean change in DBP from baseline to week 6 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -1.02, 95% CI 2-sided [-3.42 to 1.38]
Statistical Analysis 12: Comparison: Placebo vs Bexagliflozin 20 mg; Week 6: Difference in LS mean change in DBP from baseline to week 6 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.84, 95% CI 2-sided [-3.22 to 1.54]
Statistical Analysis 13: Comparison: Placebo vs Bexagliflozin 5 mg; Week 12: Difference in LS mean change in SBP from baseline to week 12 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; p = 0.3001, ANCOVA — P-value from Type III F-test; Study center, treatment, visit and a treatment-by-visit interaction as fixed effects; prior anti-diabetic treatment and baseline SBP as covariates; Difference of LS Means = -2.16, 95% CI 2-sided [-6.26 to 1.94]
Statistical Analysis 14: Comparison: Placebo vs Bexagliflozin 10 mg; Week 12: Difference in LS mean change in SBP from baseline to week 12 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; p = 0.0343, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 5, analysis 13]; Difference of LS Means = -4.41, 95% CI 2-sided [-8.49 to -0.33]
Statistical Analysis 15: Comparison: Placebo vs Bexagliflozin 20 mg; Week 12: Difference in LS mean change in SBP from baseline to week 12 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; p = 0.0679, ANCOVA; [statistical method as in outcome 5, analysis 13]; Difference of LS Means = -3.83, 95% CI 2-sided [-7.95 to 0.28]
Statistical Analysis 16: Comparison: Placebo vs Bexagliflozin 5 mg; Week 12: Difference in LS mean change in DBP from baseline to week 12 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; p = 0.0776, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 5, analysis 13]; Difference of LS Means = -2.24, 95% CI 2-sided [-4.73 to 0.25]
Statistical Analysis 17: Comparison: Placebo vs Bexagliflozin 10 mg; Week 12: Difference in LS mean change in DBP from baseline to week 12 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; p = 0.2415, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 5, analysis 13]; Difference of LS Means = -1.47, 95% CI 2-sided [-3.95 to 1.00]
Statistical Analysis 18: Comparison: Placebo vs Bexagliflozin 20 mg; Week 12: Difference in LS mean change in DBP from baseline to week 12 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; p = 0.1086, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 5, analysis 13]; Difference of LS Means = -2.04, 95% CI 2-sided [-4.54 to 0.46]

6. Secondary Outcome: Change in HbA1c Over Time
Description: The least square mean (LSM) change from baseline to Week 2, Week 6 and Week 12 was analyzed using the Mixed-Effect Model Repeated Measure (MMRM) Analysis of Covariance (ANCOVA) model using 95% Confidence Intervals (CIs) for the between-group mean changes. The LSM change was calculated by excluding HbA1c data obtained after rescue medication.
Time Frame: Baseline to Week 2, Week 6 and Week 12
Population: Only subject with a value at the specified time is included
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
Number analyzed (Participants) | 72 | 71 | 72 | 75
percentage of HbA1c
  Week 2: number analyzed (Participants) | 69 | 69 | 72 | 74
  Week 2 | -0.00 (0.04) | -0.09 (0.04) | -0.13 (0.04) | -0.13 (0.04)
  Week 6: number analyzed (Participants) | 68 | 66 | 70 | 74
  Week 6 | 0.13 (0.06) | -0.32 (0.06) | -0.36 (0.06) | -0.40 (0.06)
  Week 12: number analyzed (Participants) | 64 | 65 | 68 | 68
  Week 12 | 0.24 (0.08) | -0.31 (0.08) | -0.44 (0.08) | -0.56 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Bexagliflozin 5 mg; Week 2: Difference in LS Mean change in HbA1c (%) from baseline to Week 2 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.09, 95% CI 2-sided [-0.20 to 0.03]
Statistical Analysis 2: Comparison: Placebo vs Bexagliflozin 10 mg; Week 2: Difference in LS Mean change in HbA1c (%) from baseline to Week 2 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.13, 95% CI 2-sided [-0.24 to -0.02]
Statistical Analysis 3: Comparison: Placebo vs Bexagliflozin 20 mg; Week 2: Difference in LS Mean change in HbA1c (%) from baseline to Week 2 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.13, 95% CI 2-sided [-0.24 to -0.02]
Statistical Analysis 4: Comparison: Placebo vs Bexagliflozin 5 mg; Week 6: Difference in LS Mean change in HbA1c (%) from baseline to Week 6 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.45, 95% CI 2-sided [-0.62 to -0.28]
Statistical Analysis 5: Comparison: Placebo vs Bexagliflozin 10 mg; Week 6: Difference in LS Mean change in HbA1c (%) from baseline to Week 6 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.49, 95% CI 2-sided [-0.66 to -0.32]
Statistical Analysis 6: Comparison: Placebo vs Bexagliflozin 20 mg; Week 6: Difference in LS Mean change in HbA1c (%) from baseline to Week 6 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; Difference of LS Means = -0.53, 95% CI 2-sided [-0.70 to -0.36]
Statistical Analysis 7: Comparison: Placebo vs Bexagliflozin 5 mg; Week 12: Difference in LS Mean change in HbA1c (%) from baseline to Week 12 was obtained by comparing Bexagliflozin 5 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.55, 95% CI 2-sided [-0.76 to -0.34]
Statistical Analysis 8: Comparison: Placebo vs Bexagliflozin 10 mg; Week 12: Difference in LS Mean change in HbA1c (%) from baseline to Week 12 was obtained by comparing Bexagliflozin 10 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.68, 95% CI 2-sided [-0.89 to -0.47]
Statistical Analysis 9: Comparison: Placebo vs Bexagliflozin 20 mg; Week 12: Difference in LS Mean change in HbA1c (%) from baseline to Week 12 was obtained by comparing Bexagliflozin 20 mg group and Placebo group; Test type: Superiority; p < 0.0001, ANCOVA — P-value from Type III F-test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.80, 95% CI 2-sided [-1.01 to -0.59]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Week -12 (S2, Washout period) to Week 14 (V5, Follow up period)
Arm/Group | Placebo | Bexagliflozin 5 mg | Bexagliflozin 10 mg | Bexagliflozin 20 mg
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/72 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 3/72 | 2/76
Other Adverse Events (participants affected / at risk) | 12/72 | 15/72 | 18/72 | 17/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Bexagliflozin 5 mg (N=72) | Bexagliflozin 10 mg (N=72) | Bexagliflozin 20 mg (N=76)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=72) | Bexagliflozin 5 mg (N=72) | Bexagliflozin 10 mg (N=72) | Bexagliflozin 20 mg (N=76)
Nasopharyngitis (Infections and infestations) | 3 | 5 | 4 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 3
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has no publication right.

DOCUMENTS (2):
  • Study Protocol (2015-02-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT02390050/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT02390050/SAP_001.pdf